CLINICAL TRIAL: NCT07324993
Title: Analysis of the Effects of a 4-week Low-intensity Training With and Without Blood Flow Restriction in People With Rotator Cuff-related Shoulder Pain
Brief Title: Effects of a 4-week Low-intensity Training With Blood Flow Restriction in People With Rotator Cuff-related Shoulder Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Adrián Escriche Escuder, Assistant professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-FIS-3960959
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Related Shoulder Pain
Keywords: blood flow restriction; exercise; rotator cuff-related shoulder pain
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low resistance exercise with blood occlusion (Experimental): Eight sessions of exercise during 4 weeks, 30% repetition maximum, and 50% blood occlusion
  Interventions: Device: Resistance exercise with BFR
- Low resistance exercise without blood flow restriction (Active Comparator): Eight sessions of exercise during 4 weeks, 30% repetition maximum, without blood occlusion
  Interventions: Procedure: Resistance exercise without BFR

INTERVENTIONS:
Device: Resistance exercise with BFR — Three exercises: external rotation at 0°, internal rotation at 0° and elevation in the scapular plane. 4 sets (30, 15, 15, reps to fatigue) with a intensity of 30% RM and a 50% of arterial occlusion pressure. 30" rest between sets, 2' rest between exercises.
  Arms: Low resistance exercise with blood occlusion
Procedure: Resistance exercise without BFR — Three exercises: external rotation at 0°, internal rotation at 0° and elevation in the scapular plane. 4 sets (30, 15, 15, reps to fatigue) with a intensity of 30% RM and a without flow restriction application (cuff applied without pressure). 30" rest between sets, 2' rest between exercises.
  Arms: Low resistance exercise without blood flow restriction

SUMMARY:
This study aims to analyze the effects of 4 weeks of low-intensity exercise with and without blood flow restriction (BFR) on pain, fear of movement, catastrophizing about pain, strength, and disability in a population with rotator cuff-related shoulder pain. There are two modalities corresponding to the same exercises under different blood flow restriction conditions: 1) 3 low-intensity exercises (30% 1RM) with BFR (50% AOP); 2) 3 low-intensity exercises (30% 1RM) without BFR.

Participants will be randomly assigned to one of two groups and will undergo a 4-week intervention. The variables of interest will be assessed in each group for subsequent analysis and comparison.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65.
* Shoulder symptoms lasting at least 3 months.
* Pain in the proximal anterolateral aspect of the shoulder, aggravated by abduction.
* At least two of the following tests positive: Jobe test, resisted external rotation test, Hawkins-Kennedy test, Neer test, painful arc between 60 and 120 degrees of shoulder abduction.

Exclusion Criteria:

* Pain of an intensity that prevents performance of the proposed exercises.
* Active arm elevation less than 90 degrees.
* Clinical signs of a complete tear (positive delayed external and internal rotation sign and positive drop arm test).
* Suspected frozen shoulder (50% reduction or more than 30° loss of passive shoulder external rotation).
* Primary diagnosis of shoulder instability or acromioclavicular pathology.
* Shoulder pain due to primary involvement in the cervical or thoracic region
* Corticosteroid injection within the last 6 weeks.
* Presence of diseases such as inflammatory arthritis, neurological diseases, fibromyalgia, malignant tumors, or polymyalgia rheumatica.
* Presence of comorbidities that increase cardiovascular risk, such as hypertension, diabetes, or heart failure.
* Presence of more than one thromboembolism risk factor (obesity, history of thrombosis, prolonged immobilization, recent surgery, use of contraceptives, etc.).
* Presence of active skin lesions in the area where the sleeve will be placed, recent scars or burns, or chronic dermatological diseases that compromise skin integrity,
* Participation in upper limb exercise programs in the last month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pain intensity during movement (Visual Analogue Scale, 0-10) | Baseline, 2 weeks, and 4 weeks.
  Pain intensity perceived on a Visual Analogue Scale during movement (flexion and abduction movement without load), being 0 no pain and 10 the worst pain imaginable.

SECONDARY OUTCOMES:
Pain intensity at rest (Visual Analogue Scale, 0-10) | Baseline, 2 weeks, and 4 weeks.
  Pain intensity perceived on a Visual Analogue Scale, at rest, being 0 no pain and 10 the worst pain imaginable.
Pressure pain threshold | Before the session, immediately after, and 1 hour post-intervention
  Pressure pain threshold measured in the middle deltoid (peripheral sensitivity) and tibialis anterior (central sensitivity), using an algometer.
Kinesiophobia | Baseline, 2 weeks, and 4 weeks.
  Assessment of fear of movement or reinjury, assessed via the self-administered Tampa Scale of Kinesiophobia questionnaire.
Occurrence of adverse effects | Immediately after the intervention, 1 hour, 6 hours, 24 hours.
  Occurrence of adverse effects (e.g., pain, delayed onset muscle soreness, sudden weakness of the trained limb, redness or swelling of the trained limb, etc.) by self-report.
Pain Catastrophizing | Baseline, 2 weeks, and 4 weeks.
  Assessment of pain catastrophizing, measured using the self-report Pain Catastrophizing Scale (PCS), which evaluates exaggerated negative mental responses to actual or anticipated pain. The final score ranges from 0 to 52, with higher scores reflecting higher levels of catastrophizing.
Pain and Disability | Baseline, 2 weeks, and 4 weeks.
  Assessment of pain and disability, measured using the self-report Shoulder Pain and Disability Index (SPADI). The score ranges from 0 to 100. A score of 0 indicates best, 100 indicates worst. A higher score shows more disabillity.
Shoulder Disability | Baseline, 2 weeks, and 4 weeks.
  Assessment of shoulder disability, measured using the self-report Disabilities of the Arm, Shoulder, and Hand questionnaire (DASH). The final score ranges from 0 (no disability) to 100 (severe/maximal disability), calculated from patient-rated difficulty on a 5-point scale for 30 items, with higher scores indicating greater impairment in arm, shoulder, and hand function.
Muscle Strength | Baseline, 2 weeks, and 4 weeks.
  Assessment of supraspinatus and internal and external rotator muscle strength, measured using a strap-secured handheld dynamometer.
Satisfaction with methodology | 4 weeks.
  Assessment of participant satisfaction with the methodology used, measured at the end of the program using a 5-point scale: very satisfied (5), satisfied (4), neutral (3), dissatisfied (2), very dissatisfied (1).

CONTACTS AND LOCATIONS:
Overall Officials: Adrián Escriche-Escuder, PhD, Principal Investigator — Universitat de València

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study will be available from the corresponding author upon reasonable request.